CLINICAL TRIAL: NCT00163085
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study To Explore The Efficacy And Safety Of The NR2B NMDA Antagonist CP-101,606 In Patients With Idiopathic Parkinson's Disease
Brief Title: The Effects of an NR2B NMDA Antagonist, CP-101,606, in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A1611007
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — traxoprodil mesylate

INTERVENTIONS:
Drug: NR2B NMDA Antagonist CP-101,606 (traxoprodil)

SUMMARY:
To determine the effects of the NMDA antagonist, CP-101,606, in subjects with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* 30- 80-year-old PD patients (UK Parkinson's Disease Brain Bank criteria) with a Hoehn & Yahr stage score of 2-5 in the "off" state.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-05; Study Completion 2006-01

PRIMARY OUTCOMES:
Dyskinesia Rating Scale

SECONDARY OUTCOMES:
Fingertapping

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Portland, Oregon, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1611007&StudyName=The+Effects+of+an+NR2B+NMDA+Antagonist%2C+CP%2D101%2C606%2C+in+Patients+with+Parkinson%27s+Disease